CLINICAL TRIAL: NCT00250445
Title: A Randomized, Double-Blind, Active-Comparator-Controlled, Parallel-Group Study to Evaluate the Safety of Etoricoxib in Patients With Osteoarthritis or Rheumatoid Arthritis
Brief Title: A Study to Evaluate the Safety of an Investigational Drug (Etoricoxib) in Patients With Osteoarthritis (OA) or Rheumatoid Arthritis (RA)(0663-066)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-066; 2005_100
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Rheumatoid Arthritis,Osteoarthritis
Keywords: Arcoxia
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0663, etoricoxib
Drug: Comparator: Diclofenac sodium

SUMMARY:
The study is designed to compare the risk of cardiovascular events (heart attacks, strokes) in patients receiving either etoricoxib or diclofenac. It will also compare the gastrointestinal tolerability of the two medicines. The study will be conducted in patients with either rheumatoid or osteo-arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a clinical diagnosis of either Osteoarthritis or Rheumatoid Arthritis and in the opinion of the investigator will require chronic nonsteroidal anti-inflammatory or COX-2 inhibitor therapy for at least 1.5 years

Exclusion Criteria:

* Concurrent medical or arthritic disease that could confound or interfere with efficacy evaluation.
* Concomitant therapy of warfarin, heparin, high-dose aspirin (>100 mg/day).
* Impaired kidney function, clinical gastrointestinal malabsorption, congestive heart failure with symptoms that occur at rest, unstable angina, uncontrolled high blood pressure, active hepatitis/hepatic disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23498 (Actual)
Dates: Start 2003-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Confirmed Thrombotic Cardiovascular Serious Adverse Experiences based on combined data from this trial and MK0663 Protocols 061 & 072 (GI Tolerability in OA Patients and GI Tolerability Study in RA Patients ), respectively.

SECONDARY OUTCOMES:
Incidence of Confirmed Thrombotic Cardiovascular Serious Adverse Experiences from this trial alone. Gastrointestinal tolerability based on the percentage of patients that discontinue for clinical or laboratory gastrointestinal adverse experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Cannon CP, Curtis SP, FitzGerald GA, Krum H, Kaur A, Bolognese JA, Reicin AS, Bombardier C, Weinblatt ME, van der Heijde D, Erdmann E, Laine L; MEDAL Steering Committee. Cardiovascular outcomes with etoricoxib and diclofenac in patients with osteoarthritis and rheumatoid arthritis in the Multinational Etoricoxib and Diclofenac Arthritis Long-term (MEDAL) programme: a randomised comparison. Lancet. 2006 Nov 18;368(9549):1771-81. doi: 10.1016/S0140-6736(06)69666-9. PMID 17113426
- [Background] Laine L, Curtis SP, Cryer B, Kaur A, Cannon CP; MEDAL Steering Committee. Assessment of upper gastrointestinal safety of etoricoxib and diclofenac in patients with osteoarthritis and rheumatoid arthritis in the Multinational Etoricoxib and Diclofenac Arthritis Long-term (MEDAL) programme: a randomised comparison. Lancet. 2007 Feb 10;369(9560):465-73. doi: 10.1016/S0140-6736(07)60234-7. PMID 17292766
- [Background] Krum H, Curtis SP, Kaur A, Wang H, Smugar SS, Weir MR, Laine L, Brater DC, Cannon CP. Baseline factors associated with congestive heart failure in patients receiving etoricoxib or diclofenac: multivariate analysis of the MEDAL program. Eur J Heart Fail. 2009 Jun;11(6):542-50. doi: 10.1093/eurjhf/hfp054. Epub 2009 Apr 19. PMID 19380329
- [Background] Laine L, Curtis SP, Langman M, Jensen DM, Cryer B, Kaur A, Cannon CP. Lower gastrointestinal events in a double-blind trial of the cyclo-oxygenase-2 selective inhibitor etoricoxib and the traditional nonsteroidal anti-inflammatory drug diclofenac. Gastroenterology. 2008 Nov;135(5):1517-25. doi: 10.1053/j.gastro.2008.07.067. Epub 2008 Aug 3. PMID 18823986
- [Background] Laine L, Goldkind L, Curtis SP, Connors LG, Yanqiong Z, Cannon CP. How common is diclofenac-associated liver injury? Analysis of 17,289 arthritis patients in a long-term prospective clinical trial. Am J Gastroenterol. 2009 Feb;104(2):356-62. doi: 10.1038/ajg.2008.149. Epub 2009 Jan 27. PMID 19174782
- [Background] Combe B, Swergold G, McLay J, McCarthy T, Zerbini C, Emery P, Connors L, Kaur A, Curtis S, Laine L, Cannon CP. Cardiovascular safety and gastrointestinal tolerability of etoricoxib vs diclofenac in a randomized controlled clinical trial (The MEDAL study). Rheumatology (Oxford). 2009 Apr;48(4):425-32. doi: 10.1093/rheumatology/kep005. Epub 2009 Feb 17. PMID 19223284
- [Background] Krum H, Swergold G, Curtis SP, Kaur A, Wang H, Smugar SS, Weir MR, Laine L, Brater DC, Cannon CP. Factors associated with blood pressure changes in patients receiving diclofenac or etoricoxib: results from the MEDAL study. J Hypertens. 2009 Apr;27(4):886-93. doi: 10.1097/HJH.0b013e328325d831. PMID 19516186